CLINICAL TRIAL: NCT04990011
Title: Evaluation of Amnion Chorion Membrane in the Repair of Oro Antral Communication
Brief Title: Amnion Chorion Membrane and Oroantral Communication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: amnion chorion-2019
Record Dates: First submitted 2021-07-08; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Oroantral Communication
MeSH Terms: conditions — Oroantral Fistula

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BioXclude amnion chorion membrane (Experimental)
  Interventions: Procedure: BioXclude amnion chorion membrane

INTERVENTIONS:
Procedure: BioXclude amnion chorion membrane — The OAC will be closed by the Bioxclude ACM Amnion chorion membrane which is applied over the extraction socket then supported with a buccal advanced flap.

SUMMARY:
An oroantral communication is a relatively common yet, serious complication following the extraction of posterior maxillary teeth because of their close relationship to the maxillary sinus.

Several surgical techniques exist for the repair of oroantral communication, including local and free flaps, tissue expansion, allogenic tissue, and biomaterials.

The present study aims to evaluate the use of the BioXclude amnion chorion membrane in the repair of oroantral communication.

DETAILED DESCRIPTION:
This study will be performed on ten patients who have oroantral communication after extracting posterior maxillary teeth. The oroantral communication will be repaired by using the BioXclude amnion chorion membrane.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be free of any relevant systemic diseases.
* Patients with recent oroantral communication (O.A.C) (24:72) hours .
* Good oral hygiene

Exclusion Criteria:

* An immune compromised state.
* Previous sinus disease.
* History of sinus surgery.
* Presence of intra-antral foreign bodies and need for cold well-luc procedure.
* Presence of intra-sinus pathology

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
success of surgery | 1 month
  Surgery will be considered successful in case of negative nose-blowing 1-month postoperatively, absence of infection, absence of dehiscence or other healing complication

SECONDARY OUTCOMES:
Pain level | 12 hours
  Post-operative pain measure by patients rating 12 h after surgery using visual analogue scale (VAS) of 100 unit on three-point scale with: 0-34 as mild pain, 35 - 64 as moderate pain and 65 - 100 as severe pain
Change in bone formation | at 3rd, 6th months
  Evaluation of bone formation at the communication site by computed tomography will be measured at 3 months and 6 months post operatively

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt